CLINICAL TRIAL: NCT03452774
Title: SYNERGY-AI: Artificial Intelligence Based Precision Oncology Clinical Trial Matching and Registry
Status: Recruiting | Type: Observational
Sponsor: Massive Bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SYNERGY-AI
Record Dates: First submitted 2018-02-13; First posted 2018-03-02 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Cancer, Metastatic; Cancer; Cancer of Pancreas; Cancer of Liver; Cancer of Stomach; Cancer Liver; Cancer of Rectum; Cancer of Kidney; Cancer of Esophagus; Cancer of Cervix; Cancer of Colon; Cancer of Larynx; Cancer, Lung; Cancer, Breast; Cancer, Advanced; Cancer Prostate; Cancer of Neck; Cancer of Skin; Neuroendocrine Tumors; Carcinoma; Mismatch Repair Deficiency; BRCA Gene Rearrangement; Non Hodgkin Lymphoma; Leukemia; Non Small Cell Lung Cancer; Cholangiocarcinoma; Glioblastoma; Central Nervous System Tumor; Melanoma; Urothelial Carcinoma; Bladder Cancer; Ovarian Cancer; Endometrial Cancer; Testicular Cancer; Breast Cancer; COVID; Myelofibrosis; Myeloproliferative Neoplasm; Myeloproliferative Disorders; Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Myelodysplastic Syndromes
Keywords: artificial intelligence; virtual tumor board; clinical trial; clinical trial matching; electronic medical record; machine learning; cost of care; targeted therapy; immunotherapy; precision medicine; precision oncology; cancer; value based care; real world data; data analytics
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Rectal Neoplasms; Kidney Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Laryngeal Neoplasms; Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Head and Neck Neoplasms; Skin Neoplasms; Neuroendocrine Tumors; Carcinoma; Turcot syndrome; Lymphoma, Non-Hodgkin; Leukemia; Carcinoma, Non-Small-Cell Lung; Cholangiocarcinoma; Glioblastoma; Central Nervous System Neoplasms; Melanoma; Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Testicular Neoplasms; Primary Myelofibrosis; Myeloproliferative Disorders; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Eligible adult and pediatric pts with advanced solid and hematological malignancies, for whom the decision to consider CTE has already been made by their primary providers (PP).
  Interventions: Other: Clinical Trial Matching

INTERVENTIONS:
Other: Clinical Trial Matching — Using a proprietary application programming interface (API) linked to existing electronic health records (EHR) platforms, individual clinical data is extracted, analyzed and matched to a parametric database of existing institutional and non-institutional CT. Machine learning algorithms allow for dynamic matching based on CT allocation and availability for optimized matching.

SUMMARY:
International registry for cancer patients evaluating the feasibility and clinical utility of an Artificial Intelligence-based precision oncology clinical trial matching tool, powered by a virtual tumor boards (VTB) program, and its clinical impact on pts with advanced cancer to facilitate clinical trial enrollment (CTE), as well as the financial impact, and potential outcomes of the intervention.

DETAILED DESCRIPTION:
The SYNERGY Registry is an international prospective, observational cohort study of eligible adult and pediatric pts with advanced solid and hematological malignancies, for whom the decision to consider CTE has already been made by their primary providers (PP). Using a proprietary application programming interface (API) linked to existing electronic health records (EHR) platforms, individual clinical data is extracted, analyzed and matched to a parametric database of existing institutional and non-institutional CT. Machine learning algorithms allow for dynamic matching based on CT allocation and availability for optimized matching. Patients voluntarily enroll into the registry, which is non-interventional with no protocol-mandated tests/procedures - all treatment decisions are made at the discretion of PP in consultation with their pts, based on the AI CT matching report, and VTB support. CTE will be assessed on variables including biomarkers, barriers to enrollment. Study duration anticipated as ~36 mo (~24-mo enrollment followed by 12 mo of data collection, to occur every 3 mo). The primary analysis will be performed 12 mo after last pt enrolled. The impact time to initiation of CTE on PFS and OS will be estimated by Kaplan-Meier and Cox multivariable survival analysis. Enrollment is ongoing, with a target of ≥50,000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Pts with solid and hematological malignancies;
* Pts cancer-related biomarkers, gene variants, fusion and rearrangements (by immunohistochemistry, PCR, FISH or NGS): PD-L1, MSI (MMR), Claudin18.2, HER2/Neu, Tumor mutational burden/load (TMB), ABL1, ACVR1B, AKT1, AKT2, AKT3, ALK, APC, AR, ATM, ATRX, AURKA, AURKB, BAP1, BCL2, BCL6, BRAF, BRCA1, BRCA2, BTK, CCND1, CCND2, CCND3, CDK4, CDK6, CDKN1A/B, CEBPA, CHEK1, CHEK2, CSF1R, CTNNB1, DAXX, DDR1/2, DNMT3A, EGFR, ERBB2, ERBB3, ERBB4, ERCC4, ER, ESR1, FANCA, FAS, FBXW7, FGFR1, FGFR2, FGFR3, FGFR4, FLT3, GATA3, GATA6, GNAS, HDAC1, HGF, HRAS, IDH1, IDH2, IGF1R, JAK1, JAK2, JAK3, KDR (VEGFR2), KIT, KRAS, MAP2K2 (MEK2), MAP3K1, MCL1, MDM2, MDM4, MEN1, MET, MSH2, MSH3, MSH6, MTOR, MUTYH, MYC, MYCL (MYCL1), NF1, NF2, NOTCH1, NPM1, NRAS, NTRK1, NTRK2, NTRK3, PALB2, PARP1, PARP2, PARP3, PBRM1, PDCD1 (PD1), PDCD1LG2 (PD-L2), PDGFRA, PDGFRB, PIK3C, PMS2, POLD1, POLE, PRDM1, PTCH1, PTEN, RAF1, RB1, RET, RICTOR, ROS1, RPTOR, SDHA/B/C, SMAD, SMARC, SMO, STK11, TGFBR2, TP53, TSC1, TSC2, VEGFA, VHL, WT1, ZNF217, ZNF703, CEACAM, NRG1, among others.

These biomarkers should be determined by local laboratory, external vendor, or next generation sequencing platform

* Decision to consider clinical trial pre-screening enrollment (CTE) by primary provider and/or patient

Exclusion Criteria:

* ECOG PS > 2;
* Abnormal organ function;
* Hospice enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observational cohort study of eligible adult and pediatric pts with advanced solid and hematological malignancies, for whom the decision to consider clinical trial enrollment (CTE) has already been made by their primary providers (PP).
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2038-12 (Estimated); Study Completion 2040-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients Eligible for CTE versus Actual CTE | Through study completion, an average of 1 year
  CTE Accrual

SECONDARY OUTCOMES:
Impact of CTE on Overall Survival (OS), estimated by Kaplan-Meier and Cox multivariable survival analysis | 4 years
  OS
Impact of CTE on Progression-Free Survival (PFS), estimated by Kaplan-Meier and Cox multivariable survival analysis | 4 years
  PFS
Identification of Barriers to CTE | Through study completion, an average of 1 year
  To identify barriers to accruals to clinical trials, as measured and reported by a questionnaire
Real World Data Analytics | Through study completion, an average of 1 year
  To Analyze Individual Standard of Care Chemotherapy Utilization (nominal), across treatment lines (numeric); data will be combined and aggregated to report chemotherapy utilization rate (%).
Virtual Tumor Board Utilization | Through study completion, an average of 1 year
  VTB Use Rate
Time from Intervention to Actual CTE (months) | Through study completion, an average of 1 year
  Time to CTE

CONTACTS AND LOCATIONS:
Overall Officials: Selin Kurnaz, PhD, Principal Investigator — Massive Bio, Inc.
Locations (68):
- United States (67):
  - Massive Bio SYNERGY-AI site, Birmingham, Alabama
  - Massive Bio SYNERGY-AI site, Mobile, Alabama
  - Massive Bio SYNERGY-AI site, Scottsdale, Arizona
  - Massive Bio SYNERGY-AI site, Little Rock, Arkansas
  - Massive Bio SYNERGY-AI site, Duarte, California
  - Massive Bio SYNERGY-AI site, Irvine, California
  - Massive Bio SYNERGY-AI site, La Jolla, California
  - Massive Bio SYNERGY-AI site, Orange, California
  - Massive Bio SYNERGY-AI site, San Francisco, California
  - Massive Bio SYNERGY-AI site, Stanford, California
  - Massive Bio SYNERGY-AI site, Aurora, Colorado
  - Massive Bio SYNERGY-AI site, Denver, Colorado
  - Massive Bio SYNERGY-AI site, Littleton, Colorado
  - Massive Bio SYNERGY-AI site, Hartford, Connecticut
  - Massive Bio SYNERGY-AI site, Norwalk, Connecticut
  - Massive Bio SYNERGY-AI site, Newark, Delaware
  - Massive Bio SYNERGY-AI site, Jacksonville, Florida
  - Massive Bio SYNERGY-AI site, Miami, Florida
  - Massive Bio SYNERGY-AI site, Tampa, Florida
  - Massive Bio SYNERGY-AI site, Atlanta, Georgia
  - Massive Bio SYNERGY-AI site, Savannah, Georgia
  - Massive Bio SYNERGY-AI site, Boise, Idaho
  - Massive Bio SYNERGY-AI site, Chicago, Illinois
  - Massive Bio SYNERGY-AI site, Iowa City, Iowa
  - Massive Bio SYNERGY-AI site, New Orleans, Louisiana
  - Massive Bio SYNERGY-AI site, Scarborough, Maine
  - Massive Bio SYNERGY-AI site, Baltimore, Maryland
  - Massive Bio SYNERGY-AI site, Bethesda, Maryland
  - Massive Bio SYNERGY-AI site, Silver Spring, Maryland
  - Massive Bio SYNERGY-AI site, Towson, Maryland
  - Massive Bio SYNERGY-AI site, Worcester, Massachusetts
  - Massive Bio SYNERGY-AI site, Ann Arbor, Michigan
  - Massive Bio SYNERGY-AI site, Lansing, Michigan
  - Massive Bio SYNERGY-AI site, Duluth, Minnesota
  - Massive Bio SYNERGY-AI site, Hattiesburg, Mississippi
  - Massive Bio SYNERGY-AI site, Kansas City, Missouri
  - Massive Bio SYNERGY-AI site, St Louis, Missouri
  - Massive Bio SYNERGY-AI site, Billings, Montana
  - Massive Bio SYNERGY-AI site, Omaha, Nebraska
  - Massive Bio SYNERGY-AI site, New Brunswick, New Jersey
  - Massive Bio SYNERGY-AI site, Albuquerque, New Mexico
  - Massive Bio SYNERGY-AI site, Buffalo, New York
  - Massive Bio SYNERGY-AI site, Hempstead, New York
  - Massive Bio SYNERGY-AI site, Manhasset, New York
  - Massive Bio SYNERGY-AI site, New York, New York
  - Massive Bio SYNERGY-AI site, Staten Island, New York
  - Massive Bio SYNERGY-AI site, Chapel Hill, North Carolina
  - Massive Bio SYNERGY-AI site, Winston-Salem, North Carolina
  - Massive Bio SYNERGY-AI site, Fargo, North Dakota
  - Massive Bio SYNERGY-AI site, Cincinnati, Ohio
  - Massive Bio SYNERGY-AI site, Columbus, Ohio
  - Massive Bio SYNERGY-AI site, Mayfield Heights, Ohio
  - Massive Bio SYNERGY-AI site, Tulsa, Oklahoma
  - Massive Bio SYNERGY-AI site, Portland, Oregon
  - Massive Bio SYNERGY-AI site, Philadelphia, Pennsylvania
  - Massive Bio SYNERGY-AI site, Providence, Rhode Island
  - Massive Bio SYNERGY-AI site, Greenville, South Carolina
  - Massive Bio SYNERGY-AI site, Memphis, Tennessee
  - Massive Bio SYNERGY-AI site, Nashville, Tennessee
  - Massive Bio SYNERGY-AI site, Dallas, Texas
  - Massive Bio SYNERGY-AI site, Houston, Texas
  - Massive Bio SYNERGY-AI site, Temple, Texas
  - Massive Bio SYNERGY-AI site, Salt Lake City, Utah
  - Massive Bio SYNERGY-AI site, Charlottesville, Virginia
  - Massive Bio SYNERGY-AI site, Seattle, Washington
  - Massive Bio SYNERGY-AI site, Morgantown, West Virginia
  - Massive Bio SYNERGY-AI site, Milwaukee, Wisconsin
- Massive Bio SYNERGY-AI site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No